CLINICAL TRIAL: NCT05337462
Title: Étude Pilote du Séquençage Rapide du génome Humain Des Patients sévèrement Malades Dans Les Soins Intensifs en pédiatrie
Brief Title: Pilot Study of Rapid Whole Genome Sequencing of Severely Ill Patients in Pediatric Intensive Care in Belgium
Acronym: rWGS_v3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, AIME LUMAKA, Doctor, Centre Hospitalier Universitaire de Liege
Other Study IDs: 2020/143
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Rare Diseases
Keywords: Rare Diseases; Whole Genome Sequencing
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Remaining DNA samples are stored in the Biobank fo the University Hospitals of Liège.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multi-site, non-randomized (single arm) study to evaluate the feasibility, the yield and clinical utility of trio WGS in 30 critically ill patients in neonatology intensive care units (NICU) and pediatric intensive care units (PICU) in Belgium. Results are expected to be returned within 7 days after receipt of blood samples in the laboratory. Primary outcome will be evaluated after clinical interpretation, whereas secondary outcome will be evaluated from the clinical utility survey to be completed by clinical geneticists.

DETAILED DESCRIPTION:
This is a prospective, multi-site, non-randomized (single arm) study to evaluate the feasibility, the yield and clinical utility of trio WGS in critically ill patients in neonatology intensive care units (NICU) and pediatric intensive care units (PICU) in Belgium. Each proband responding to our eligibility criteria will receive a trio WGS.

Blood samples from enrolled probands and their parents will be collected and shipped to the Laboratoire de Génétique Humaine, University of Liège, Liège, Belgium, which is a research facility. Blood samples will be lysed using the Illumina Lysis Kit. Lysis product will be used for library preparation with Illumina DNA PCR-Free Prep, Tagmentation library preparation kit and IDT® for Illumina® DNA/RNA Unique Dual Indexes Set A, Tagmentation. Pooled libraries will be sequenced on a NovaSeq 6000. Sequencing data will be automatically transferred to Cloud Space (BaseSpace Sequence Hub) were primary bioinformatic analysis will be performed upon completion of sequencing and data transfer. Annotated variant calling files for SNVs and CNVs will be analyzed with Moon (Invitae) and in-house bioinformatic analysis solutions. Clinical interpretation will be performed by the principal investigator.

WGS results were communicated to pediatrician. The clinical utility survey was filled by clinical geneticists at least a month after the return of sequencing results.

ELIGIBILITY:
Inclusion Criteria:

* at least two major malformations involving two different systems
* A specific malformation highly suggestive of a genetic etiology, including but not limited to any of the following abnormalities:

  * Choanal atresia,
  * Coloboma,
  * Hirschsprung's disease,
  * Meconium ileus (except in case of prematurity),
  * Agenesis of the corpus callosum or Lissencephaly
* An abnormal laboratory test suggesting a genetic disease or a complex metabolic phenotype, including but not limited to any of the following:

  * Conventional abnormal neonatal screening
  * Conjugated hyperbilirubinemia not due to total parental nutrition (TPN) cholestasis
  * Hyperammonemia
  * Lactic acidosis not due to poor perfusion
  * Refractory or severe hypoglycaemia
* An abnormal response to standard treatment for a major underlying condition

  * Significant hypotonia
  * Persistent seizures
* Infant with high-risk stratification on assessment of a Brief Resolved Unexplained Event (BRUE) with any of the following features :

  * Recurrent events without respiratory infection
  * Recurrent seizures observed
  * Unexplained cardiopulmonary resuscitation (CPR) required
  * Significantly abnormal biochemical status, including but not limited to electrolytes, bicarbonate or lactic acid, venous blood gases, glucose, or other tests suggestive of an inborn error of metabolism
* Significantly abnormal electrocardiogram (ECG), including but not limited to possible channelopathies, arrhythmias, cardiomyopathies, myocarditis, or structural heart disease
* Positive family history of:

  * Arrhythmia
  * BRUE at the brother
  * Developmental delay / mental retardation
  * Inborn error of metabolism or genetic disease without genetic diagnosis
  * Long QT Syndrome (LQTS)
  * Sudden unexplained death (including unexplained car accident or drowning) in first- or second-degree relatives before age 35, and especially as an infant.

Exclusion Criteria:

* An infection with a normal response to treatment
* A confirmed genetic diagnosis explaining the disease
* Hypoxic ischemic encephalopathy (HIE) with a clear precipitating event
* Isolated prematurity
* Isolated transient tachypnea of the newborn (TTN)
* Isolated unconjugated hyperbilirubinemia
* Non-viable neonates
* Entity of multifactorial cause or unknown genetic cause, including but not limited to any of the following: Sequence of amniotic bands, Isolated Pierre Robin sequence, Spina bifida

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All critically ill newborns of pediatric patients admitted in intensive care units of the participating institutions during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 7 days
  # of molecular diagnostic / total # of probands in percentage
Turn-around time | One week
  The average time (in hours) from the sample reception in the laboratory to the electronic signature of the test report.

SECONDARY OUTCOMES:
Correlation with clinical diagnostic | one week
  Percentage of clinical diagnostic confirmed by the WGS testing
Guidance to disease management | One month after the results are returned
  Percentage of patients in whom the disease management plan was adjusted based on the results of the WGS

CONTACTS AND LOCATIONS:
Overall Officials: AIME LUMAKA, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (2):
- Belgium (2):
  - Centre Hospitalier Régional de la Citadelle, Liège
  - CHC Mont-Légia, Liège

IPD SHARING:
Plan to Share IPD: No
Deidentified and curated variant and limited phenotype information will be submitted to ClinVar. ClinVar is a freely accessible, public archive of reports of the relationships between human genomic variations and clinical phenotypes hosted by the National Center for Biotechnology Information (NCBI) and funded by Intramural National Institutes of Health (NIH) funding. No personal health information (PHI) or information identifying the participant or family will be submitted.